CLINICAL TRIAL: NCT01886989
Title: Postprandial Effects of Polyphenol-rich Cocoa Beverage on Glucose, Insulin, Lipids, Oxidative Stress and Inflammation in Type 2 Diabetic Patients
Brief Title: Cocoa Polyphenols and Postprandial Metabolism in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arpita Basu (Other)
Responsible Party: Sponsor-Investigator, Arpita Basu, Associate Professor, Oklahoma State University
Organization: Oklahoma State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HE-12-52
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; cocoa polyphenols; postprandial glycemia; postprandial lipemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cocoa (Experimental): Cocoa polyphenols (960mg)
  Interventions: Dietary Supplement: Cocoa polyphenols
- Placebo (Placebo Comparator): Placebo powder (109mg polyphenols) in water
  Interventions: Dietary Supplement: Cocoa polyphenols

INTERVENTIONS:
Dietary Supplement: Cocoa polyphenols — Cocoa polyphenols (960mg) reconstituted in water

SUMMARY:
This study aims to investigate the postprandial effects of cocoa supplementation in glucose and lipids, and surrogate markers of atherosclerosis in patients with type 2 diabetes. The investigators aim to test the hypothesis that cocoa will lower high-fat mixed meal breakfast-induced postprandial rise of glucose, lipids and markers of atherosclerosis in patients with diabetes. Randomized cross-over controlled trial, in which participants will be assigned to the placebo or cocoa group with breakfast meal. Patients with type 2 diabetes(n=25) will qualify for the study. The participants will be asked to consume 2 cups cocoa or placebo beverage on 2 separate postprandial study days. Both groups will receive high-fat mixed meal breakfast on each day. Blood draws and blood pressure (including HDI) measurements will be conducted at fasting, 30 min, 1,2, 4 & 6 hours postprandial each day for 2 days.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of type 2diabetes

Exclusion Criteria:

* on insulin therapy

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure (mm Hg) | 2.5 years
  Change in blood pressure and vascular function following cocoa and placebo intervention

SECONDARY OUTCOMES:
Glucose (mg/dL) | 2.5 years
  Change in glucose levels at fasting, 30min, 1, 2, 4, & 6 hours postprandial following cocoa and placebo intervention
Blood lipids | 2.5 years
  Change in lipids and lipoprotein levels at fasting, 30min, 1, 2, 4, & 6 hours postprandial following cocoa
Inflammation | 2.5 years
  Change in CRP and interleukins levels at fasting, 30min, 1, 2, 4, & 6 hours postprandial following cocoa

CONTACTS AND LOCATIONS:
Overall Officials: ARPITA BASU, PHD, Principal Investigator — Oklahoma State University
Locations (1):
- Department of Nutritional Sciences, Stillwater, Oklahoma, United States

REFERENCES:
- [Derived] Davis DW, Tallent R, Navalta JW, Salazar A, Lyons TJ, Basu A. Effects of Acute Cocoa Supplementation on Postprandial Apolipoproteins, Lipoprotein Subclasses, and Inflammatory Biomarkers in Adults with Type 2 Diabetes after a High-Fat Meal. Nutrients. 2020 Jun 27;12(7):1902. doi: 10.3390/nu12071902. PMID 32605005
- [Derived] Basu A, Betts NM, Leyva MJ, Fu D, Aston CE, Lyons TJ. Acute Cocoa Supplementation Increases Postprandial HDL Cholesterol and Insulin in Obese Adults with Type 2 Diabetes after Consumption of a High-Fat Breakfast. J Nutr. 2015 Oct;145(10):2325-32. doi: 10.3945/jn.115.215772. Epub 2015 Sep 2. PMID 26338890